CLINICAL TRIAL: NCT01394601
Title: RECONNECT-S ALPHA: A Non-interventional Study to Observe Real-life Allocation of Antipsychotics in the Acute Inpatient Management of Schizophrenia
Brief Title: A Study to Observe Real-life Allocation of Antipsychotics in Acute Inpatient Management of Schizophrenia
Acronym: RECONNECT-S
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NRU-ATC-2011/1
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Schizophrenia
Keywords: Antipsychotics; schizophrenia; acute inpatient
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Clinical Practice
Oversight: Data Monitoring Committee: No

SUMMARY:
RECONNECT-S ALPHA is a multicentre study to observe the management of schizophrenic patients who are hospitalized due to an acutely agitated psychotic episode. The patients should be managed according to normal clinical practice until discharge time. Data will be collected by review of medical records of the hospitalisation prior the study visit. During the study the patients will conduct one visit on the day of their discharge after hospitalisation due to an acutely agitated psychotic episode. On the study visit data on demographics, diagnosis and medical history will be recorded. Data on antipsychotic and concomitant medication will be collected by review of medical records.

DETAILED DESCRIPTION:
RECONNECT-S ALPHA: A non-interventional study to observe real-life allocation of antipsychotics in the acute inpatient management of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* male or female patients,
* 18 years or older,
* meeting the diagnostic criteria for schizophrenia stated in The Diagnostic and Statistical Manual of Mental Disorders,
* meeting 4th edition (DSM-IV) criteria hospitalization due to an acutely agitated psychotic episode.

Exclusion Criteria:

* patient in acutely agitated state upon discharge from the hospital,
* current participation in any clinical trial,
* previous enrolment in the present NIS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical Practice
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients using of atypical antipsychotics.Daily dosage of atypical antipsychotics Mode of administration of atypical antipsychotics. | up to 6 months

SECONDARY OUTCOMES:
Treatment with of only one antipsychotic during the hospitalization.Use of psychometric scales to evaluate the disease symptoms. Relationship between the patient characteristics and the use of antipsychotic during hospitalisation and after discharge | up to 6 months
Number of antipsychotics used during the hospitalization due to an acutely agitated psychotic episode. Use of treatment concomitant to antipsychotics during the hospitalization | up to 6 months
Relationship between medication used during the hospitalization and prescribed as maintenance antipsychotic medication upon discharge. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Study Director — AstraZeneca; Nikolay Govorin, Principal Investigator — Chita State Medical Akademy of Roszdraw
Locations (8):
- Russia (8):
  - Research Site, Chita
  - Research Site, Ivanovo
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Clinical Site, Novosibirsk
  - Clinical Site, S-Petersburg
  - Research Site, Samara
  - Research Site, Yekaterinburg